CLINICAL TRIAL: NCT01000909
Title: Venous Pressure Measurement of the Great Saphenous Vein Using Controlled Compression Ultrasound in Healthy Persons and Patients With Chronic Venous Disease as a New Non Invasive Method for Investigation of the Pathophysiology in Primary Varicose Veins
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Christoph Thalhammer, MD, USZ
Other Study IDs: CT-02-2009-USZ
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Venous Insufficiency
MeSH Terms: interventions — High-Energy Shock Waves; Venous Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Ultrasound (venous pressure measurement) — increased venous pressure is predictive for chronic venous insufficiency

SUMMARY:
Part I:

Proof of concept trial to achieve normal venous pressure values under different provocation maneuvers in healthy persons

Part II:

Non invasive measurement of venous pressure under different provocation maneuvers in patients with chronic venous disease

ELIGIBILITY:
Inclusion criteria:

Part I:

* Healthy persons without clinical signs of venous disease, informed consent

Part II:

* Patients with chronic venous disease with complete incompetence of the great saphenous vein (Hach IV)
* Informed consent

Exclusion criteria:

Part I:

* Clinical signs of venous disease, former deep vein thrombosis (DVT)

Part II:

* Former deep vein thrombosis, former vein surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic venous disease with complete incompetence of the great saphenous vein
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-07; Study Completion 2010-07

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland